CLINICAL TRIAL: NCT00307749
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled, 24-Week Dose Finding Study to Evaluate the Efficacy and Safety of 20mg, 40mg and 80mg of MCC-257 in Patients With Mild to Moderate Diabetic Polyneuropathy
Brief Title: Safety and Efficacy of MCC-257 in the Treatment of Diabetic Polyneuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MCC-257-A03
Record Dates: First submitted 2006-03-27; First posted 2006-03-28 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Diabetic Polyneuropathy
Keywords: Neuropathy; Nerve Conduction
MeSH Terms: conditions — Diabetic Neuropathies | interventions — MCC-257

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: MCC-257
- 3 (Experimental)
  Interventions: Drug: MCC-257
- 4 (Experimental)
  Interventions: Drug: MCC-257

INTERVENTIONS:
Drug: Placebo — once daily for 24 weeks
  Arms: 1
Drug: MCC-257 — 20mg, once daily for 24 weeks
  Arms: 2
Drug: MCC-257 — 40mg, once daily for 24 weeks
  Arms: 3
Drug: MCC-257 — 80mg, once daily for 24 weeks
  Arms: 4

SUMMARY:
The primary objectives of the study are to evaluate the efficacy and safety of three doses of MCC-257 in patients with mild to moderate diabetic polyneuropathy

DETAILED DESCRIPTION:
The study will use a double-blind, randomized, placebo-controlled, fixed-dose, parallel-group design. Patients will be randomized equally to 1 of 4 treatment groups: MCC-257 20 mg, MCC-257 40 mg, MCC-257 80 mg, or placebo, given once daily for 24 weeks. The study will consist of 2 periods: 1) a screening period of up to 21 days prior to baseline, including a formal screening visit; and 2) a 24-week treatment period, during which patients will take the study treatment, and have various assessments performed during 4 visits.

ELIGIBILITY:
Inclusion Criteria:

* The patient is male or female, 18-70 years of age
* The patient has either type 1 or type 2 diabetes
* The patient has mild to moderate diabetic neuropathy
* The patient is free from other clinically significant illness or disease, as determined by medical history, physical examination, laboratory evaluations, and other safety tests

Exclusion Criteria:

* Being treated with anticoagulants other than aspirin, such as warfarin, digoxin, Plavix
* BMI>40
* A significant disorder or a condition other than diabetes that can cause symptoms or physical conditions that mimic peripheral neuropathy or interfere with cognition
* Any proximal neuropathy, clinically evident nerve entrapment, or any focal trauma potentially affecting nerve function
* Women of childbearing potential who do not refrain from sexual activity or use adequate contraception
* Pregnant or lactating women
* An ALT or AST value >2X upper limit of normal (ULN)
* Clinically significant cardiovascular disease within the last six (6) months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2006-03; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Nerve Conduction Studies | Day 1, Week 24

SECONDARY OUTCOMES:
Nerve fiber density | Day 1, Week 24
QST | Day 1, Week 12, Week 24
Symptom | Day 1, Week 12, Week 24
Clinical Global Impression | Week 12, Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Professor, Principal Investigator — Information at Mitsubishi Pharma America